CLINICAL TRIAL: NCT06490653
Title: Comparison of the Efficacy of Tranexamic Acid and Blood Stopper Treatments in Bleeding Control in Patients With Epistaxis: A Randomized Controlled Trial
Brief Title: Tranexamic Acid Versus Blood Stopper Treatments in Epistaxis Management
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Şeref Kerem Çorbacıoğlu, Emergency Medicine Department, Ankara Ataturk Sanatorium Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0048
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Epistaxis Nosebleed
Keywords: Epistaxis; Nosebleed; Ankaferd; Tranexamic acid
MeSH Terms: conditions — Epistaxis | interventions — ankaferd blood stopper

STUDY DESIGN:
Intervention Model Description: In this study, there are two parallel treatment arms (tranexamic acid and blood stopper (Ankaferd®) determined by randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was designed so that patients and researchers in all roles (care provider, outcome assessor, and statistician) were masked to the treatment arms. Following the enrolment, the principal investigator will be contacted to find out which treatment arm the patient will be enrolled in according to the predetermined order. According to the assigned treatment arm, the relevant treatment will be prepared by another researcher in a physically non-distinguishable. A care provider will administer the prepared treatment and assess whether bleeding has stopped approximately 10 minutes after administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): Patients will be asked to clean their nose with tap water as part of the routine treatment before the administration. After then, Tranexamic acid (500mg/5 ml) will be sprayed through the bleeding side nostril and then external pressure will be applied to the nose for 10 minutes.
  Interventions: Drug: Blood Stopper (Ankaferd)
- Blood Stopper (Ankaferd) (Experimental): Patients will be asked to clean their noses with tap water as part of the routine treatment before the administration. After then, 5 ml of Ankaferd® will be sprayed through the bleeding side nostril and external nasal pressure will be performed for 10 minutes.
  Interventions: Drug: Blood Stopper (Ankaferd)

INTERVENTIONS:
Drug: Blood Stopper (Ankaferd) — 5 ml of Ankaferd® will be sprayed through the bleeding side nostril and external nasal pressure will be performed for 10 minutes.

SUMMARY:
In this randonmized controlled trial, aim to compare the effectiveness of local administration of tranexamic acid and blood stopper (Ankaferd®) on cessation of bleeding in epistaxis patients.

DETAILED DESCRIPTION:
Anterior tamponade is frequently used in the management of anterior epistaxis. However, this procedure is often uncomfortable for patients. Therefore, instead of this physical tampon, various pharmacologic agents such as tranexamic acid, blood stoppers (ankaferd®), and adrenaline can be used in epistaxis management. Although the superiority of various agents used in the management of anterior epistaxis has been evaluated in published network meta-analyses, these meta-analyses do not compare ankaferd and Tranexamic acid since there are no studies with each other. In order to close the gap in the existing literature, this study aims to evaluate the superiority of local administration of tranexamic acid and ankaferd® in terms of cessation of bleeding in patients with anterior epistaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with epistaxis will present to the emergency department with non-traumatic epistaxis and whose bleeding do not stop with simple external compression for 10 minutes.

Exclusion Criteria:

* Patients demonstrating hemodynamic instability
* Patients with documented allergy to tranexamic acid or Ankaferd
* patients with known bleeding disorders,
* patients using anticoagulants,
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cessation of bleeding | 10-minutes after performing local drug interventions.
  Primary outcome was definition cessation in bleeding at 10-minutes after performing local drug interventions.

SECONDARY OUTCOMES:
Re-bleeding | From cessation of bleeding to re-bleeding within 24-hours.
  The secondary outcome was a comparison of the re-bleeding rate within 24 hours in the two treatments groups.

IPD SHARING:
Plan to Share IPD: No